CLINICAL TRIAL: NCT04393168
Title: Proof-of-concept Interventional Study to Evaluate the Feasibility of the New Method, LymphMonitor 1.0, to Assess Lymphatic Function, Consisting of Indocyanine Green-based Lymphatic Specific Tracer. and a Custom Fluorescence Measuring Investigational Device LymphMeter 1.0.
Brief Title: Proof-of-concept Study of LymphMonitor 1.0 to Assess the Lymphatic Vessel Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nicole Lindenblatt (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Zurich University of Applied Sciences (Other); University Hospital, Zürich (Other); NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor-Investigator, Nicole Lindenblatt, Deputy Director of the Division of Plastic and Hand Surgery, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POCLymphMonitor 1.0; 2019-01823 (Registry Identifier: SNCTP clinical trials registry)
Record Dates: First submitted 2020-05-09; First posted 2020-05-19 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Lymphedema; Secondary Lymphedema
Keywords: lymphedema; secondary lymphedema; fluorescence; indocyanine green
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with unilateral arm or leg lymphedema (Experimental)
  Interventions: Combination Product: Lymphatic clearance measurement

INTERVENTIONS:
Combination Product: Lymphatic clearance measurement — The indocyanine green in 5% human albumin solution (tracer) (50 μL) will be injected intradermally in both forearms or both lower legs using MicronJet600 microneedles paying attention to the contralateral symmetry of the injections. The signal at the injection sites will be measured over time using a hand-held portable device LymphMeter 1.0 for the total duration of 3 h. In the first hour, the signal will be measured every 15 minutes followed by measurements every half an hour. Immediately after injection (t=0 h), 1.5 h and 3 h after injection the skin area occupied by the tracer will be measured using a standard near-infrared camera, Fluobeam. The dermal reaction at the injection site will be assessed by observations for presence of redness/erythema and measuring its extent according to the needs. The patient will be constantly observed for the signs of allergic reactions, skin irritations or intolerances.

SUMMARY:
Lymphedema is the consequence of injured lymphatic system and is characterized by chronic, often disabling swelling of am affected body part, often arm or leg. In the western world secondary lymphedema arises most commonly after removal lymph nodes in an operation as a part of cancer treatment (for example from the armpits or the groin region), however it may also develop as a result of radiation, any other operation, infection or injury that destroys a part of lymphatic system. The disease often develops even years after the event. While there is no cure for lymphedema at present, early detection would ensure timely physiotherapy and application of compression garments that significantly slow down or stop the progression of the disease. However, presently used methods of that are used for diagnosis and evaluating the stage of the disease, are either invasive and expensive or inaccurate and can only be performed at specialized medical centres.

Therefore, we developed a simple, affordable and accurate technology, LymphMonitor 1.0 that can allow for testing how efficiently the lymphatic system is functioning. The test can be performed at the local medical centre or potentially even at home.

In this study, we investigate whether LymphMonitor 1.0 technology can distinguish between a healthy and a diseased lymphatic system (in lymphedema). This method may allow early diagnosis of lymphedema so that the development of the disease can be detected and prevented early enough. By participating in the study the lymphedema patients are making an important contribution to increasing the quality of life of lymphedema patients. In LymphMonitor 1.0 method method, a solution of a safe fluorescent dye, indocyanine green, is injected painlessly using tiny microneedles, MicronJet600TM, directly into the skin of the arm or leg. After injection, this dye is removed from the skin only through the lymphatic vessels. The intensity of the fluorescence signal corresponds to the amount of dye left in the skin. The decrease in the fluorescence signal after the injection is measured on the surface on the skin using a new device, LymphMeter 1.0. The faster the dye (and that fluorescence signal) disappears from the surface of the skin, the better the lymphatic system works. Therefore in the arm or leg affected by lymphedema the fluorescence signal will decrease much slower compared to the healthy one.

ELIGIBILITY:
Inclusion criteria:

* informed consent as documented by signature
* females and males 18 - 75 years old,
* established (stage 2 or higher) unilateral secondary arm or leg lymphedema resulting from lymphadectonomy, radiation or any other surgical treatment, infection or injury.
* good general health status.

Exclusion criteria:

* critical illness (active cancer, renal failure, hepatic dysfunction)
* active infection
* blood vascular malformations or diseases
* scleroderma
* primary lymphedema
* patients who underwent any surgical procedures for treatment of lymphedema (e.g. lymphovenous anastomosis, liposuction, lymph node transfer).
* contraindications to use ICG (VERDYE), i.e.
* patients with hypersensitivity to ICG or to sodium iodide
* patients with hypersensitivity to iodine,
* patients with hyper-thyroidism, patients with autonomic thyroid adenomas
* patients in which the injection of VERDYE was poorly tolerated in the past it must not be used again, since severe anaphylactic reactions might occur.
* hypersensitivity to albumin or its excipients
* women, who are pregnant (pregnancy test will be performed in case of women who did not undergo menopause),
* women who are breast feeding ,
* enrolment of the investigator, his/her family members, employees and other dependent persons,
* known or suspected non-compliance, drug or alcohol abuse,
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* participation in another study with investigational drug within the 30 days preceding and during the present study,
* previous enrolment into the current study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Areas under the normalized clearance curves (AUCs) | Fluorescence values measured immediately after injection and 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours after injection.
  Areas under the normalized clearance curves (AUCs) in healthy and lymphedema limbs measured over 3 hours after injection. To obtain the clearance curve, the fluorescence intensity values at the injection sites in healthy and lymphedema extremities at pre-determined timepoints

SECONDARY OUTCOMES:
other clearance parameters: clearance constant (k) and half-life of clearance (t1/2); (healthy versus diseased). | Fluorescence values measured immediately after injection and 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours after injection.
Correlation/no correlation of clearance parameters with the extent of the swelling (limb volume) in lymphedema patients. | 3 hours
dimensions of the injected dye depot measured by FluoBeam | Dimensions will be measured immediately after injection and 1.5 hours and 3 hours after injection.
  Images of the injection site over time will be recorded using Fluobeam at different and analysed.

OTHER OUTCOMES:
Safety outcomes | 3 hours
  Specific safety outcomes in this study will consist of any signs of potential allergic reactions and irritation of injection sites or any other intolerances
Safety outcomes | Through the study completion, an average of 5 hours
  Any adverse effects (AEs) and serious adverse effects (SAEs) (expected and unexpected will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Lindenblatt, M.D, PhD, Principal Investigator — University Hostpial Zurich
Locations (1):
- University Hostpial Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided